CLINICAL TRIAL: NCT00359983
Title: A Study to Evaluate the Long-term Antibody Persistence at 1, 3 & 5 Years After the Administration of a Fourth Dose of Hib-MenCY-TT Vaccine Compared to ActHIB in Subjects Boosted in a Previous Study.
Brief Title: Long-Term Antibody Persistence at 1, 3 and 5 Years After a Fourth Dose of GSK Biologicals' Hib-MenCY-TT Vaccine Compared to ActHIB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107824; 107826 (Other: GSK); 107829 (Other: GSK); NCT00360113 (obsolete NCT alias); NCT00360165 (obsolete NCT alias)
Record Dates: First submitted 2006-07-31; First posted 2006-08-03 (Estimated); Results first posted 2012-07-20 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-11

CONDITIONS: Neisseria Meningitidis; Haemophilus Influenzae Type b
Keywords: Humans; Meningococcal vaccines; Immunogenicity; Vaccines; H. influenzae type b vaccine; Conjugate; Toddlers; Comparative study; Neisseria meningitidis
MeSH Terms: conditions — Haemophilus Infections | interventions — Hib-MenCY-TT vaccine; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate

ARMS (3):
- MenHibrix 4-dose group (Experimental): Subjects received in the primary study (NCT00129129) 3 doses of MenHibrix co-administered with Pediarix and Prevnar and a 4th dose of MenHibrix co-administered with Prevnar. No vaccines were administered during this long-term persistence study.
  Interventions: Biological: MenHibrix (Hib-MenCY-TT)
- ActHIB 4-dose group (Active Comparator): Subjects received in the primary study (NCT00129129) 3 doses of ActHIB co-administered with Pediarix and Prevnar and a 4th dose of ActHIB co-administered with Prevnar. No vaccines were administered during this long-term persistence study.
  Interventions: Biological: Hib conjugate vaccine (ActHIB)
- ActHIB 3-dose + MenHibrix 4th-dose group (Experimental): Subjects received in the primary study (NCT00129129) 3 doses of ActHIB co-administered with Pediarix and Prevnar and a dose of MenHibrix co-administered with Prevnar. No vaccines were administered during this long-term persistence study.
  Interventions: Biological: MenHibrix (Hib-MenCY-TT); Biological: Hib conjugate vaccine (ActHIB)

INTERVENTIONS:
Biological: MenHibrix (Hib-MenCY-TT) — First three doses: 3 intramuscular doses Fourth dose: 1 intramuscular dose
  Other Names: GSK biologicals' Hib-MenCY-TT
  Arms: ActHIB 3-dose + MenHibrix 4th-dose group; MenHibrix 4-dose group
Biological: Hib conjugate vaccine (ActHIB) — First three doses: 3 intramuscular doses Fourth dose: 1 intramuscular dose
  Other Names: ActHIB
  Arms: ActHIB 3-dose + MenHibrix 4th-dose group; ActHIB 4-dose group

SUMMARY:
This study is evaluating antibody persistence at 1, 3 & 5 years post-fourth dose (i.e., at 2, 4 & 6 years of age, respectively) in subjects vaccinated in a previous study.

This protocol posting deals with objectives & outcome measures of the extension phase at years 1, 3 and 5. The objectives & outcome measures of the first four doses are presented in a separate protocol posting (NCT00129129).

This protocol posting has been amended in order to comply with the FDA Amendment Act of September 26, 2007.

DETAILED DESCRIPTION:
In this long-term follow-up study, no new subjects will be recruited. All subjects participating in this long-term follow-up study should have already participated in a previous study. No vaccine will be administered during the persistence phase of the study.

This Protocol Posting has been updated following Protocol amendment 3, September 2009.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female children who completed the previous four dose vaccination series study (NCT00129129). The age of the child at the 3 post-fourth dose timelines are as follows:

  * Year 1: 22 to 36 months of age.
  * Year 3: 44 to 60 months of age.
  * Year 5: 5 years post-dose 4 +/- 8 weeks
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study
* Having completed the fourth dose vaccination of study Hib-MenCY-TT-005/006

Exclusion Criteria:

Children should not have:

* received more than 4 doses of Hib or meningococcal serogroup C and Y vaccine
* had a history of H. influenzae type b, meningococcal serogroup C and Y diseases

Ages: 22 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 270 (Actual)
Dates: Start 2006-09; Primary Completion 2007-11 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (18):
- United States (18):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Waukee, Iowa
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Pittsford, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Boardman, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Greenville, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bryant KA, Marshall GS. Haemophilus influenzae type b-Neisseria meningitidis serogroups C and Y tetanus toxoid conjugate vaccine for infants and toddlers. Expert Rev Vaccines. 2011 Jul;10(7):941-50. doi: 10.1586/erv.11.90. PMID 21806393
- [Background] Marshall GS, Marchant CD, Blatter M, Aris E, Boutriau D, Poolman JT, Friedland LR, Miller JM. Immune response and one-year antibody persistence after a fourth dose of a novel Haemophilus influenzae type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine (HibMenCY) at 12 to 15 months of age. Pediatr Infect Dis J. 2010 May;29(5):469-71. doi: 10.1097/INF.0b013e3181cdd379. PMID 20072077
- [Background] Marshall GS et al. Antibody persistence 5 years after the fourth dose of a US-licensed Heamophilus influenzae type B and Neisseria meningitidis serogroups C and Y tetanus toxoid (HIBMENCY-TT) conjugate vaccine. Abstract presented at the 50th Annual Meeting of the Infectious Diseases Society of America - (IDSA-IDWeek), San Diego, 17-21 October 2012.
- [Background] Marshall GS et al. Persistence of Immunity three years after an Investigational Haemophilus influenzae type b and Neisseria meningitidis Serogroups C and Y Tetanus Toxoid (HibMenCY-TT) Conjugate Vaccine. Abstract presented at the 45th National Immunization Conference (NIC). Washington, D.C, USA, 28-31 March 2011.
- [Derived] Marshall GS, Blatter M, Marchant C, Aris E, Mesaros N, Miller JM. Antibody persistence for up to 5 years after a fourth dose of Haemophilus influenzae type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine (HibMenCY-TT) given at 12-15 months of age. Pediatr Infect Dis J. 2013 Jun;32(6):662-8. doi: 10.1097/INF.0b013e3182840e35. PMID 23340564
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 107824 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107824 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107824 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107824 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107824 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107824 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Year 1 Persistence Follow-up
Arm/Group | MenHibrix 4-dose Group | ActHIB 4-dose Group | ActHIB 3-dose + MenHibrix 4th-dose Group
Started | 138 | 70 | 62
Completed | 138 | 70 | 62
Not Completed | 0 | 0 | 0
Period: Year 3 Persistence Follow-up
Arm/Group | MenHibrix 4-dose Group | ActHIB 4-dose Group | ActHIB 3-dose + MenHibrix 4th-dose Group
Started | 103 | 47 | 51
Completed | 103 | 47 | 51
Not Completed | 0 | 0 | 0
Period: Year 5 Persistence Follow-up
Arm/Group | MenHibrix 4-dose Group | ActHIB 4-dose Group | ActHIB 3-dose + MenHibrix 4th-dose Group
Started | 95 | 44 | 42
Completed | 95 | 44 | 42
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenHibrix 4-dose Group | ActHIB 4-dose Group | ActHIB 3-dose + MenHibrix 4th-dose Group | Total
Number analyzed (Participants) | 138 | 70 | 62 | 270
Age, Continuous [Mean (Standard Deviation); unit: Months]
  Months | 27.4 (3.37) | 28.2 (4.05) | 28.4 (3.69) | 27.8 (3.64)
Gender [Count of Participants; unit: Participants]
  Female | 67 | 35 | 33 | 135
  Male | 71 | 35 | 29 | 135

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti- Polyribosylribitol Phosphate (Anti-PRP) Antibody Concentrations Greater Than or Equal to 0.15 Microgram Per Milliliter
Description: Results up to 5 years after the fourth dose are presented.
Time Frame: One year, three years, and five years after the fourth dose vaccination.
Population: Analysis was done on the ATP cohort for persistence of each respective timepoint in all evaluable subjects who had assay results available for at least one tested antigen and who had a blood sample taken between 309 and 645 days (Year 1 data), 1039 and 1375 days (Year 3 data) and 1770 and 1882 days (Year 5 data) after administration of fourth dose.
Measure: Number; unit: Subjects
Arm/Group | MenHibrix 4-dose Group | ActHIB 4-dose Group | ActHIB 3-dose + MenHibrix 4th-dose Group
Number analyzed (Participants) | 116 | 51 | 46
Subjects
  Year 1 (N=116; 51; 46) | 116 | 49 | 46
  Year 3 (N=61; 28; 36) | 60 | 26 | 36
  Year 5 (N=84; 39; 37) | 83 | 36 | 36

2. Primary Outcome: Number of Subjects With Neisseria Meningitidis Serogroup C (MenC) Antibody Titers Greater Than or Equal to 1:8 as Measured by Serum Bactericidal Assay Using Human Complement (hSBA)
Description: Results up to 5 years after the fourth dose are presented.
Time Frame: One year, three years, and five years after the fourth dose vaccination.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | MenHibrix 4-dose Group | ActHIB 4-dose Group | ActHIB 3-dose + MenHibrix 4th-dose Group
Number analyzed (Participants) | 116 | 52 | 48
Subjects
  Year 1 (N=116; 52; 48) | 112 | 12 | 34
  Year 3 (N=59; 27; 35) | 48 | 3 | 20
  Year 5 (N=76; 38; 34) | 63 | 8 | 25

3. Primary Outcome: Number of Subjects With Neisseria Meningitidis Serogroup Y (MenY) Antibody Titers Greater Than or Equal to 1:8 as Measured by Serum Bactericidal Assay Using Human Complement (hSBA)
Description: Results up to 5 years after the fourth dose are presented.
Time Frame: One year, three years, and five years after the fourth dose vaccination.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | MenHibrix 4-dose Group | ActHIB 4-dose Group | ActHIB 3-dose + MenHibrix 4th-dose Group
Number analyzed (Participants) | 105 | 50 | 47
Subjects
  Year 1 (N=105; 50; 47) | 88 | 0 | 31
  Year 3 (N=58; 26; 34) | 39 | 4 | 19
  Year 5 (N=82; 38; 35) | 57 | 7 | 19

4. Secondary Outcome: Anti-PRP Geometric Mean Concentrations (GMCs)
Description: Concentration were measured as Geometric Mean Concentrations expressed as microgram per milliliter (µg/mL).
  Results up to 5 years after the fourth dose are presented.
Time Frame: One year, three years, and five years after the fourth dose vaccination.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | MenHibrix 4-dose Group | ActHIB 4-dose Group | ActHIB 3-dose + MenHibrix 4th-dose Group
Number analyzed (Participants) | 116 | 51 | 46
µg/mL
  Year 1 (N=116; 51; 46) | 2.400 [1.937 to 2.975] | 1.943 [1.308 to 2.887] | 1.162 [0.808 to 1.672]
  Year 3 (N=61; 28; 36) | 1.169 [0.851 to 1.605] | 1.031 [0.625 to 1.700] | 0.898 [0.623 to 1.293]
  Year 5 (N=84; 39; 37) | 1.248 [0.970 to 1.605] | 0.803 [0.524 to 1.231] | 0.689 [0.447 to 1.064]

5. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations Greater Than or Equal to 1.0 Microgram Per Milliliter
Description: Results up to 5 years after the fourth dose are presented.
Time Frame: One year, three years, and five years after the fourth dose vaccination.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | MenHibrix 4-dose Group | ActHIB 4-dose Group | ActHIB 3-dose + MenHibrix 4th-dose Group
Number analyzed (Participants) | 116 | 51 | 46
Subjects
  Year 1 (N= 116; 51; 46) | 88 | 35 | 24
  Year 3 (N=61; 28; 36) | 33 | 14 | 14
  Year 5 (N= 84; 39; 37) | 47 | 17 | 10

6. Secondary Outcome: hSBA-MenC Geometric Mean Titers (GMTs)
Description: Titers are given as Geometric Mean Titers as measured by human serum bactericidal assay (hSBA) and expressed as the reciprocal of the dilution resulting in 50% inhibition.
  Results up to 5 years after the fourth dose are presented.
Time Frame: One year, three years, and five years after the fourth dose vaccination.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MenHibrix 4-dose Group | ActHIB 4-dose Group | ActHIB 3-dose + MenHibrix 4th-dose Group
Number analyzed (Participants) | 116 | 52 | 48
Titer
  Year 1 (N= 116; 52; 48) | 150.1 [116.5 to 193.4] | 3.9 [2.7 to 5.5] | 26.3 [14.8 to 46.5]
  Year 3 (N= 59; 27; 35) | 41.9 [25.8 to 68.0] | 2.7 [1.9 to 3.7] | 16.0 [7.4 to 34.9]
  Year 5 (N= 76; 38; 34) | 69.8 [41.8 to 116.5] | 3.6 [2.4 to 5.4] | 44.2 [18.8 to 103.9]

7. Secondary Outcome: Number of Subjects With hSBA-MenC Titers Greater Than or Equal to 1:4
Description: Results up to 5 years after the fourth dose are presented.
Time Frame: One year, three years, and five years after the fourth dose vaccination.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | MenHibrix 4-dose Group | ActHIB 4-dose Group | ActHIB 3-dose + MenHibrix 4th-dose Group
Number analyzed (Participants) | 116 | 52 | 48
Subjects
  Year 1 (N= 116; 52; 48) | 112 | 12 | 34
  Year 3 (N= 59; 27; 35) | 48 | 3 | 20
  Year 5 (N= 76; 38; 34) | 63 | 8 | 26

8. Secondary Outcome: hSBA-MenY Geometric Mean Titers (GMTs)
Description: as for outcome 6
Time Frame: One year, three years, and five years after the fourth dose vaccination.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MenHibrix 4-dose Group | ActHIB 4-dose Group | ActHIB 3-dose + MenHibrix 4th-dose Group
Number analyzed (Participants) | 105 | 50 | 47
Titer
  Year 1 (N= 105; 50; 47) | 128.8 [86.2 to 192.5] | 2.0 [2.0 to 2.0] | 41.1 [20.4 to 82.9]
  Year 3 (N= 58; 26; 34) | 29.9 [16.9 to 52.8] | 3.5 [2.0 to 6.3] | 16.6 [8.0 to 34.4]
  Year 5 (N= 82; 38; 35) | 26.8 [17.7 to 40.4] | 3.6 [2.4 to 5.5] | 17.8 [8.4 to 37.7]

9. Secondary Outcome: Number of Subjects With hSBA-MenY Titers Greater Than or Equal to 1:4
Description: Results up to 5 years after the fourth dose are presented.
Time Frame: One year, three years, and five years after the fourth dose vaccination.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | MenHibrix 4-dose Group | ActHIB 4-dose Group | ActHIB 3-dose + MenHibrix 4th-dose Group
Number analyzed (Participants) | 105 | 50 | 47
Subjects
  Year 1 (N= 105; 50; 47) | 89 | 0 | 31
  Year 3 (N= 58; 26; 34) | 39 | 4 | 19
  Year 5 (N= 82; 38; 35) | 57 | 7 | 19

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed in subjects for Year 1, Year 3 and Year 5 respectively.
Description: No information on other frequent adverse events was collected during this study. Only information on serious adverse events assessed by the investigator as causally related to the vaccination was collected.
Arm/Group | MenHibrix 4-dose Group | ActHIB 4-dose Group | ActHIB 3-dose + MenHibrix 4th-dose Group
Serious Adverse Events (participants affected / at risk) | 0/138 | 0/70 | 0/62
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.